CLINICAL TRIAL: NCT00955305
Title: A Phase II Randomized Trial of Paclitaxel, Carboplatin, Bevacizumab With or Without IMC-A12 in Patients With Advanced Non-squamous, Non-small Cell Lung Cancer
Brief Title: Paclitaxel, Carboplatin, and Bevacizumab With or Without Cixutumumab in Treating Patients With Stage IV or Recurrent Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed to accrual due to the end of the clinical development program with cixutumumab.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01960; NCI-2011-01960 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E3508 (Other: ECOG-ACRIN Cancer Research Group); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Results first posted 2016-09-08 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Large Cell Lung Carcinoma; Lung Adenocarcinoma; Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer; Bronchioloalveolar Lung Carcinoma
Keywords: Non-Small Cell Lung Cancer; cixutumumab
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; cixutumumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (CPB) (Active Comparator): Patients receive carboplatin intravenously (IV) over 30 minutes, paclitaxel IV over 3 hours, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Treatment with bevacizumab may continue in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel
- Arm B (CPB+cixutumumab) (Experimental): Patients receive carboplatin, paclitaxel, and bevacizumab as in Arm A. Patients also receive cixutumumab (IMC-A12) IV over 1 hour on days 1, 8, and 15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Treatment with bevacizumab and cixutumumab may continue in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Biological: Cixutumumab; Drug: Paclitaxel

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: NSC 704865; Avastin; rhuMAb-VEGF
Drug: Carboplatin — Given IV
  Other Names: CBDCA; Paraplatin; JM-8; NSC 241240
Biological: Cixutumumab — Given IV
  Other Names: NSC 742460; IMC-A12
  Arms: Arm B (CPB+cixutumumab)
Drug: Paclitaxel — Given IV
  Other Names: Taxol

SUMMARY:
This randomized phase II trial studies how well carboplatin, paclitaxel, and bevacizumab (CPB) work when given with or without cixutumumab in treating patients with non-small cell lung cancer that is stage IV or has come back (recurrent). Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Other types of monoclonal antibodies, such as cixutumumab, may find tumor cells and help kill them. It is not yet known whether giving more than one drug (combination chemotherapy) together with bevacizumab is more effective when given with or without cixutumumab in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression-free survival with the combination of carboplatin, paclitaxel, and bevacizumab, and +/- IMC-A12 (cixutumumab) in patients with advanced, non-squamous, non-small cell lung cancer.

SECONDARY OBJECTIVES:

I. To evaluate overall survival and response rate of the above combination in patients with non-squamous, advanced non-small cell lung cancer.

II. To evaluate the toxicities of the above combination in patients with non-squamous advanced non-small cell lung cancer.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A (CPB): Patients receive carboplatin intravenously (IV) over 30 minutes, paclitaxel IV over 3 hours, and bevacizumab IV over 30-90 minutes on day 1.

ARM B (CPB+cixutumumab): Patients receive carboplatin, paclitaxel, and bevacizumab as in Arm A. Patients also receive cixutumumab (IMC-A12) IV over 1 hour on days 1, 8, and 15.

In both arms, treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Treatment with bevacizumab and cixutumumab may continue in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed with non-squamous, non-small cell lung cancer (NSCLC)
* Advanced NSCLC defined as either recurrent disease after prior radiation or surgery or stage IV (M1a or M1b) based on the TNM staging system (American Joint Committee on Cancer [AJCC] 2009)
* Measurable disease as defined by the revised Response Evaluation Criteria in Solid Tumors (RECIST version 1.1). All sites of disease (of target and non-target disease sites) must be obtained within 4 weeks prior to randomization
* A head computed tomography (CT) or magnetic resonance imaging (MRI) required within 4 weeks prior to randomization
* Prior radiation therapy (RT) is allowed if it has been completed 3 weeks prior to randomization and patient has recovered from any adverse events related to RT
* Brain metastases are allowed, provided they have been treated with surgery and/or radiotherapy, the patient is neurologically stable, and repeat brain imaging shows no progression in the brain; at least 6 weeks should have elapsed from the time of craniotomy and at least 4 weeks from radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) ≥ 1500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin within institutional upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 x ULN
* Fasting blood glucose within normal range (fasting < 120 mg/dL or below ULN)
* Alkaline phosphatase (ALP) ≤ 3 x ULN
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN
* Urine dipstick must be ≤ 0-1+ within 2 weeks (14 days) of randomization; if urine dipstick result is > 1+, a calculation of urine protein creatinine (UPC) ratio is required; patients must have a UPC ratio < 1.0 to participate in the study
* Neuropathy, if present at baseline, must be ≤ Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Patients with a history of hypertension must be well-controlled (≤ 150/90) on a stable regimen of anti-hypertensive therapy
* Women of childbearing potential and sexually active males should use an accepted and effective method of contraception while on treatment and for 3 months thereafter

Exclusion Criteria:

* Prior chemotherapy or biologic/molecular targeted therapy for advanced NSCLC. Prior chemotherapy and/or biological/molecular targeted therapy as part of initial potentially curative therapy (one regimen of induction and/or adjuvant and/or concurrent chemoradiotherapy) was allowed provided it had been completed 1 year or more prior to randomization
* Prior treatment with IMC-A12 or another insulin-like growth factor 1 receptor (IGF-1R) inhibitor
* Patients on therapeutic anticoagulation; patient's international normalized ratio (INR) must be ≤ 1.5 or partial thromboplastin time (PTT) ≤ upper limits of normal within 2 weeks prior to randomization to be eligible; prophylactic anticoagulation of venous access devices is allowed provided the above criteria have been met
* Prior allergic reaction to compounds of chemical or biologic composition similar to those of IMC-A12
* Hypersensitivity to any component of bevacizumab
* Poorly controlled diabetes mellitus
* History of other invasive malignancies unless there is no active disease and all treatment has been completed ≥ 3 years prior to randomization; patients with history of in-situ malignancies and curatively resected nonmelanomatous skin cancer are eligible
* History of thrombotic or hemorrhagic disorders
* History of bleeding diathesis or coagulopathy
* ≥ grade 2 bleeding or any bleeding requiring intervention within 4 weeks prior to randomization
* History of gross hemoptysis (defined as ≥ 1/2 teaspoon of bright red blood)
* Any of the following within 6 months prior to randomization:

  * Abdominal fistula
  * Gastrointestinal perforation
  * Intra-abdominal abscess
  * Previous myocardial infarction
  * History of any central nervous system (CNS) cerebrovascular ischemia
  * New York Heart Association (NYHA) > class II congestive heart failure or severe heart failure
  * Unstable or symptomatic angina pectoris
  * History of stroke
  * Significant vascular disease
  * Symptomatic peripheral vascular disease
* Ongoing, serious cardiac arrhythmia requiring medication at time of randomization
* Ongoing, active infection or ongoing fever at the time of randomization or any co-existing medical condition, psychiatric illness or limitations that would interfere with compliance of study requirements
* History of hypertensive crisis or hypertensive encephalopathy
* Any of the following within 4 weeks prior to randomization: a serious non-healing wound, ulcer, bone fracture, or major surgical procedure
* Anticipated major surgical procedure(s) during the course of the study
* Receiving daily treatment with aspirin (> 325 mg/day) or non-steroidal anti-inflammatory agents (NSAIDs) known to inhibit platelet function for chronic conditions; patients must not be receiving treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix), and/or cilostazol (Pletal); if patient was receiving any of the following: aspirin (> 325 mg/day), NSAID, and/or anti-platelet drugs, patient must have discontinued its use ≥ 1 week prior to randomization
* Pregnant or breast-feeding
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2010-03; Primary Completion 2016-01 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios (Ethan) Argiris, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (165):
- United States (165):
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Charlotte Hungerford Hospital Center for Cancer Care, Torrington, Connecticut
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Hospital, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - PinnacleHealth Cancer Center-Community Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Dallas VA Medical Center, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - West Virginia University Charleston, Charleston, West Virginia
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Argiris, A., Lee, J., Leach, J.W., Schiller, J.H.: Safety analysis of a phase II randomized trial of carboplatin (C), Paclitaxel (P), bevacizumab (B) with or without cixutumumab (CX) in patients (pts) with advanced non-squamous, non-small cell lung cancer (NSCLC). J Clin Oncol 2014;31(15s). Abstract e19018.
- [Derived] Argiris A, Lee JW, Stevenson J, Sulecki MG, Hugec V, Choong NW, Saltzman JN, Song W, Hansen RM, Evans TL, Ramalingam SS, Schiller JH. Phase II randomized trial of carboplatin, paclitaxel, bevacizumab with or without cixutumumab (IMC-A12) in patients with advanced non-squamous, non-small-cell lung cancer: a trial of the ECOG-ACRIN Cancer Research Group (E3508). Ann Oncol. 2017 Dec 1;28(12):3037-3043. doi: 10.1093/annonc/mdx534. PMID 28950351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to accrual on March 9, 2010 and was suspended on February 24, 2011 for safety evaluation. As the safety criterion was met, this study reopened on May 16, 2011 and closed to accrual on June 28, 2013 due to the end of the clinical development program with cixutumumab (IMC-A12) with final accrual of 175 patients.
Period: Overall Study
Arm/Group | Arm A (CPB) | Arm B (CPB+Cixutumumab)
Started | 88 | 87
Treated | 83 | 82
Eligible and Treated | 78 | 75
Completed | 0 (Treatment continued until disease progression or unacceptable toxicities.) | 0 (Treatment continued until disease progression or unacceptable toxicities.)
Not Completed | 88 | 87
Not completed — Disease progression | 39 | 41
Not completed — Adverse Event | 22 | 22
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Alternative therapy | 4 | 0
Not completed — Other complicating disease | 2 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Continued presence of residual disease | 0 | 1
Not completed — Functional decline | 2 | 0
Not completed — Maximum response achieved | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — No off-treatment reason submitted | 1 | 0
Not completed — Never started protocol treatment | 5 | 5
Not completed — Ineligible | 5 | 7

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (CPB) | Arm B (CPB+Cixutumumab) | Total
Number analyzed (Participants) | 78 | 75 | 153
Age, Continuous [Median (Full Range); unit: years] | 64 [38 to 82] | 61 [28 to 82] | 63 [28 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 38 | 35 | 73

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to progression or death without documentation of progression. For cases without progression, follow-up was censored at the date of last disease assessment without progression, unless death occurs within 3 months following the date last known progression-free, in which case the death was counted as a failure.
  Progression was evaluated using RECIST 1.1 criteria and defined as:
  1. At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm.
     OR
  2. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry; every 6 months if patient is 2 - 5 years from study entry; up to 5 years
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (CPB) | Arm B (CPB+Cixutumumab)
Number analyzed (Participants) | 78 | 75
months | 5.8 [5.4 to 7.1] | 7.0 [5.7 to 7.6]
Statistical Analysis 1: Comparison: Arm A (CPB) vs Arm B (CPB+Cixutumumab); Test type: Superiority or Other; p = 0.33, Log Rank — one-sided p-value using stratified logrank test stratified on the randomization stratification factors; Stratified log rank test stratified on the randomization stratification factors

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to death or date last known alive.
Time Frame: as for outcome 1
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (CPB) | Arm B (CPB+Cixutumumab)
Number analyzed (Participants) | 78 | 75
months | 16.2 [9.9 to 18.6] | 16.1 [12.3 to 19.4]
Statistical Analysis 1: Comparison: Arm A (CPB) vs Arm B (CPB+Cixutumumab); Test type: Superiority or Other; p = 0.95, Log Rank — two-sided p-value by stratified log rank test stratified on the randomization stratification factors; Stratified log rank test stratified on the randomization stratification factors

3. Secondary Outcome: Proportion of Patients With Objective Response
Description: Objective response was evaluated using the RECIST 1.1 criteria.
  Objective response includes complete response (CR) and partial response (PR). Objective response is defined as disappearance of all target lesions or at least a 30% decrease in the sum of the diameters of target lesions. In addition, non-target lesions do not meet the criteria for disease progression and no new lesions were observed.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry and every 6 months if patient is 2-5 years from study entry; up to 5 years
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (CPB) | Arm B (CPB+Cixutumumab)
Number analyzed (Participants) | 78 | 75
Proportion of participants | 0.462 [0.348 to 0.578] | 0.587 [0.467 to 0.699]
Statistical Analysis 1: Comparison: Arm A (CPB) vs Arm B (CPB+Cixutumumab); Test type: Superiority or Other; p = 0.15, Fisher Exact — two sided p-value by Fisher's exact test

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Description: Patients received a maximum of 6 cycles of chemotherapy and remained on bevacizumab (Arm A) or bevacizumab + cixutumumab (Arm B) continuously until evidence of documented progressive disease or unacceptable toxicity.
Arm/Group | Arm A (CPB) | Arm B (CPB+Cixutumumab)
Serious Adverse Events (participants affected / at risk) | 58/83 | 74/82
Other Adverse Events (participants affected / at risk) | 80/83 | 78/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (CPB) (N=83) | Arm B (CPB+Cixutumumab) (N=82)
Anemia (Blood and lymphatic system disorders) | 6 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 7
Fatigue (General disorders) | 5 | 17
Fever (General disorders) | 1 | 2
Infusion related reaction (General disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 9
Oral pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 6
Catheter related infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Gum infection (Infections and infestations) | 0 | 1
Joint infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 3
Mucosal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 9 | 9
Neutrophil count decreased (Investigations) | 27 | 45
Platelet count decreased (Investigations) | 8 | 21
Serum amylase increased (Investigations) | 0 | 1
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 4 | 16
Anorexia (Metabolism and nutrition disorders) | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 4 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal and connective - Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4
Reversible posterior leukoencephalopathy (Nervous system disorders) | 0 | 1
Spasticity (Nervous system disorders) | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 1 | 0
Blurred vision (Eye disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory thoracic mediastinal - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 4
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0
Hypertension (Vascular disorders) | 12 | 17
Hypotension (Vascular disorders) | 2 | 1
Thromboembolic event (Vascular disorders) | 7 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (CPB) (N=83) | Arm B (CPB+Cixutumumab) (N=82)
Anemia (Blood and lymphatic system disorders) | 64 | 58
Chills (General disorders) | 3 | 7
Edema limbs (General disorders) | 5 | 2
Fatigue (General disorders) | 66 | 69
Fever (General disorders) | 5 | 4
Infusion related reaction (General disorders) | 0 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 60 | 48
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 13
Abdominal pain (Gastrointestinal disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 27 | 25
Diarrhea (Gastrointestinal disorders) | 18 | 31
Mucositis oral (Gastrointestinal disorders) | 7 | 21
Nausea (Gastrointestinal disorders) | 38 | 49
Oral hemorrhage (Gastrointestinal disorders) | 3 | 5
Oral pain (Gastrointestinal disorders) | 5 | 12
Vomiting (Gastrointestinal disorders) | 18 | 24
Mucosal infection (Infections and infestations) | 0 | 5
Alanine aminotransferase increased (Investigations) | 10 | 14
Alkaline phosphatase increased (Investigations) | 12 | 15
Aspartate aminotransferase increased (Investigations) | 11 | 18
Creatinine increased (Investigations) | 7 | 15
Lymphocyte count decreased (Investigations) | 28 | 26
Neutrophil count decreased (Investigations) | 27 | 23
Platelet count decreased (Investigations) | 40 | 52
Weight loss (Investigations) | 19 | 35
White blood cell decreased (Investigations) | 21 | 26
Anorexia (Metabolism and nutrition disorders) | 35 | 48
Dehydration (Metabolism and nutrition disorders) | 4 | 6
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 15 | 45
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 10
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 7
Hypokalemia (Metabolism and nutrition disorders) | 6 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 9 | 7
Hyponatremia (Metabolism and nutrition disorders) | 14 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 17
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 16 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 11
Dizziness (Nervous system disorders) | 7 | 8
Dysgeusia (Nervous system disorders) | 11 | 17
Headache (Nervous system disorders) | 7 | 17
Peripheral motor neuropathy (Nervous system disorders) | 5 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 54 | 47
Blurred vision (Eye disorders) | 2 | 6
Insomnia (Psychiatric disorders) | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 37
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Hematuria (Renal and urinary disorders) | 6 | 4
Proteinuria (Renal and urinary disorders) | 21 | 17
Hypertension (Vascular disorders) | 30 | 31
Hypotension (Vascular disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less